CLINICAL TRIAL: NCT06222060
Title: Evaluation of Young Parents' Knowledge of Shaken Baby Syndrome in Maternity Wards
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN462023/CHUSTE
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-01

CONDITIONS: Shaken Baby Syndrome
Keywords: Shaken Baby Syndrome; Child abuse; Parental knowledge
MeSH Terms: conditions — Shaken Baby Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parents: Couples of parents of newborns
  Interventions: Other: Questionnaire about Shaken Baby Syndrome

INTERVENTIONS:
Other: Questionnaire about Shaken Baby Syndrome — Knowledge assessment questionnaire completed in the maternity ward by both parents

SUMMARY:
As part of everyday clinical practice, messages about preventing Shaken Baby Syndrome are delivered to young parents in maternity wards. The modality of these messages changes regularly. For example, in the near future, the messages will be delivered by video in addition to the usual practice. The investigators are setting up a prospective observational cohort study in order to evaluate and then monitor the state of knowledge of young parents on shaken baby syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Parents of newborns in maternity wards

Exclusion Criteria:

* Single parent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents of newborns in maternity wards
Sampling Method: Non-Probability Sample
Enrollment: 686 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Shaken Baby Syndrome Knowledge | Week 1, 6
  Change in the proportion of correct knowledge about Shaken Baby Syndrome : a higher level of knowledge indicates a better result.

CONTACTS AND LOCATIONS:
Overall Officials: Aymeric CANTAIS, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No